CLINICAL TRIAL: NCT04445610
Title: Measles Vaccine: Is There a Protective Role in COVID 19 Pandemic?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Al Balakosy, Tropical Medicine Department. Ain Shams University, Ain Shams University
Other Study IDs: FMASU P31a/ 2020
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus (COVID-19)
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: mild
- B: moderate
- C: severe

SUMMARY:
The following two mechanisms that explain the ability of measles vaccine to cause partial protection against COVID-19. The first is that measles vaccine may increase the ability of the immune system to fight off pathogens other than measles due to the generated bystander immunity that would enhance the overall immunity against the new coronavirus. The second is that SARS-CoV-2 is proven to have structure similarities with measles, which may cause cross-reactivity and immunity between measles vaccines and COVID-19, leading to partial protection against COVID-19 in vaccinated subjects

DETAILED DESCRIPTION:
Objectives:

1. To identify Measles IgG titre in SARS-COV2 infected patients .
2. correlate level of Measles IgG titre with the clinical severity of COVID-19 disease.

Secondary Objective To find an association of the postulated protective role of measles vaccine and SARS-COV2 infection

Criteria:

Inclusion criteria:included patients would be divided into 3 groups according to clinical severity of COVID-19 disease (mild ,moderate & severe)

* All patients with confirmed COVID 19 confirmed by positive PCR . .
* Any age or gender.

Exclusion criteria:

- Any patient refusing to be involved in the study.

Methods:

* Informed consent will be taken from each subject
* Full clinical examination.
* Evaluation of Measles Antibody Titer:

The measles virus IgG antibody titer will be determined quantitatively by ELISA for quantitative determination of IgG class antibodies against Measles virus in human serum or plasma (citrate, heparin).

- Anonymous data will be retrieved from the admitted patients' files, such as:

* CBC, CRP, AST, ALT, ESR, Serum ferritin & SARS CoV 2 RNA PCR swab results.
* Chest X ray and/or CT chest.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed COVID 19.
* Any age or gender

Exclusion Criteria:

* - Any patient refusing to be involved in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with confirmed COVID-19 presented to Ain Shams Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Viral clearance | 6 months
  Achievement of two consecutive negative PCR results for COVID 19 and discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Amira Al Balakosy, M.D, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No